CLINICAL TRIAL: NCT00619775
Title: Carotid Revascularization With ev3 Arterial Technology Evolution (CREATE) Trial
Acronym: CREATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-1007
Record Dates: First submitted 2008-02-07; First posted 2008-02-21 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2008-12

CONDITIONS: Carotid Artery Disease
Keywords: Carotid Artery Disease; Embolic Protection
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: PROTÉGÉ® GPS™ and PROTÉGÉ® RX Carotid Stent Systems and Spider Embolic Protection Device — Carotid artery stenting with distal embolic protection.

SUMMARY:
Evaluate the safety and efficacy of the Protege Stent and Spider Device in the treatment of common and/or internal carotid artery stenoses for subjects that are high risk for carotid endarterectomy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* informed consent
* for female subjects, not pregnant or planning on becoming pregnant
* meet protocol defined anatomical or clinical high risk criteria

Exclusion Criteria:

* participation in another clincial study which may affect either the pre-procedure or follow-up results
* prior stenting of the ipsilateral carotid artery
* life expectancy less than twelve months
* known allergy or intolerance of study medications or device materials
* must not meet general or angiographic exclusion criteria as defined in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2004-04; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Myocardial infarction, ipsilateral cerebrovascular accident, procedure-related contralateral CVA or death within 30 days of implantation; and ipsilateral CVA from 31 days to 1 year post-implantation | 30 days and one year

SECONDARY OUTCOMES:
Ipsilateral CVA, procedure-related contralateral CVA or death with 30 days of implantation; and ipsilateral CVA from 31 days to 1 year post-implantation | 30 days and one year
Target lesion revascularization | one year
Target vessel revascularization | one year
Primary patency at one year (<70% stenosis as measured by duplex scan) | one year
Technical success (defined as the ability to deploy the filter, place the stent over the filter wire, and recapture the filter with the resulting residual stenosis <50%) | at implant

CONTACTS AND LOCATIONS:
Overall Officials: Robert Safian, MD, Principal Investigator — Corewell Health East
Locations (31):
- United States (31):
  - Banner Baywood Heart Hospital, Mesa, Arizona
  - Scripps Memorial Hospital, La Jolla, California
  - El Camino Hospital, Mountain View, California
  - Hoag Memorial Hospital, Newport Beach, California
  - Salinas Valley Memorial Healthcare System, Salinas, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - St. Francis Medical Center, Peoria, Illinois
  - St. Vincent Hospital & Health Care Centers, Indianapolis, Indiana
  - The Heart Center of Indiana, Indianapolis, Indiana
  - Kramer & Crouse Cardiology, Shawnee Mission, Kansas
  - Terrebonne General Hospital, Houma, Louisiana
  - Southwest Medical Center, Lafayette, Louisiana
  - Union Memorial Hospital, Baltimore, Maryland
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Oakwood Hospital, Dearborn, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Louis University Medical Center, St Louis, Missouri
  - University of Buffalo Millard Fillmore Hospital, Buffalo, New York
  - Duke University Medical Center, Raleigh, North Carolina
  - Wake Heart Associates, Raleigh, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist, Columbus, Ohio
  - Holy Spirit Hospital, Harrisburg, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Pinnacle Health at Harrisburg Hospital, Wormleysburg, Pennsylvania
  - Greenville Hospital System, Greenville, South Carolina
  - Avera Heart Hospital of South Dakota, Sioux Falls, South Dakota
  - Baptist Heart Institute, Knoxville, Tennessee
  - University of Virginia, Charlottesville, Virginia
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- [Result] Safian RD, Bresnahan JF, Jaff MR, Foster M, Bacharach JM, Maini B, Turco M, Myla S, Eles G, Ansel GM; CREATE Pivotal Trial Investigators. Protected carotid stenting in high-risk patients with severe carotid artery stenosis. J Am Coll Cardiol. 2006 Jun 20;47(12):2384-9. doi: 10.1016/j.jacc.2005.12.076. PMID 16781363
- [Result] Safian RD, Bacharach JM, Ansel GM, Criado FJ. Carotid stenting with a new system for distal embolic protection and stenting in high-risk patients: the carotid revascularization with ev3 arterial technology evolution (CREATE) feasibility trial. Catheter Cardiovasc Interv. 2004 Sep;63(1):1-6. doi: 10.1002/ccd.20155. PMID 15343559